CLINICAL TRIAL: NCT05880550
Title: Response of Menstrual Irregularity and Infertility- Related Stress to Ultrasound Cavitation Combined With Aerobic Exercise in PCOS: Double Blinded Randomized Controlled Trial
Brief Title: PCOS and US Cavitation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Marwa Shafiek Mustafa Saleh, assistance professor doctor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: US cavitation and PCOS
Record Dates: First submitted 2023-05-19; First posted 2023-05-30 (Actual); Last update posted 2024-05-14 (Actual); Status verified 2024-05

CONDITIONS: PCOS (Polycystic Ovary Syndrome) of Bilateral Ovaries
MeSH Terms: conditions — Polycystic Ovary Syndrome | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- study group (Experimental)
  Interventions: Other: ultrasound cavitation in addition to aerobic ex
- control group (Active Comparator)
  Interventions: Other: aerobic exercises.

INTERVENTIONS:
Other: ultrasound cavitation in addition to aerobic ex — Ultrasonic cavitation was turned on, the program of cavitation 40 kHz was chosen, the time was adjusted at 30 minutes. The cavitational head was moved very slowly on each abdominal segment in a small circular movement for 5 minutes. After finishing the focused ultrasound of the 6 segments of the abdomen, the skin was cleaned with cotton.
  in addition to that the patients will receive aerobic exercises for 40 minutes.
  Arms: study group
Other: aerobic exercises. — the patients will do aerobic training for 40 minutes on a bicycle ergometer.
  Arms: control group

SUMMARY:
Polycystic ovary syndrome (PCOS) is the most common endocrine disorder in women of reproductive age. Women with this syndrome may have infrequent menstrual periods or amenorrhea and excess androgen levels. The ovaries develop numerous small follicles and fail to ovulate on a regular basis, with subsequent subfertility in those women that wish to conceive. Recent research stated that interventions aiming to improve QoL among infertile women with PCOS should focus on alleviating infertility-related stress, especially among women with high BMI. So, the purpose of this study is to investigate the effect of ultrasound cavitation combined with aerobic exercise on menstrual irregularity and infertility related stress in women having PCOS.

ELIGIBILITY:
Inclusion Criteria

All women in this study will be on the following criteria:

* Their ages will range from 20-35 years.
* They will be diagnosed with PCOS by Gynecologist.
* Doesn't receive any treatment for menstrual regularity and fertility during the study.
* BMI above 25kg/m²and less than 35kg/m².
* Waist /hip ratio <.88.

Exclusion Criteria

Women will be excluded if they have one of the following criteria:

* Skin diseases that prevent the application of cavitation.
* Severe cardiovascular disease.
* Other endocrine disordered (hypothyroidism hyperprolactinemia).
* Patients that who take hormonal treatment within the last 3 months before the study.

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2023-05-25 (Actual); Primary Completion 2023-08-25 (Actual); Study Completion 2023-09-25 (Actual)

PRIMARY OUTCOMES:
Infertily related Stress level | change from base line at 12 weeks.
  Infertility-Related Stress Scale is a concise, reliable, and validated tool; it facilitates quick screening for infertility's impact on intrapersonal and interpersonal life domains. The IRSS consists of 12 items rated from 1 ("no stress") to 7 ("high stress")., with higher grades means higher stress.
cortisol level | change from base line at 12 weeks.
  Saliva samples will be collected with study participants sitting upright in a comfortable position and tilting the head forward, allowing the saliva to pool on the floor of the mouth

SECONDARY OUTCOMES:
Anthrometric measurement (body mass index and waist-hip ratio) | change from base line at 12 weeks.
  BMI and waist/hip ratio Measurements of body mass index in which the weight in kilograms divided by the square of the heights in meters and waist to hip circumference measured with a soft tape at the level of the umbilicus and the anterior superior iliac spine with woman in the standing position, were made before treatment and after the end of the study period
Hormonal profile | change from base line at 12 weeks.
  Blood samples will be drown from an antecubital vein of each patient in the study on two occasions, firstly at the end at 2 nd or 3 rd day of the menstrual cycle after an overnight fasting just before starting her treatment regimen and secondly after 3 months of the treatment. It will be centrifuged within 2 hours after withdrawal. Serum will be stared at -20OC and assayed for LH and FSH with chemiluminescent enzyme immunoassay kits. Assays for fasting insulin by RIA kits and SHBG will be determined by using an immunoradiometric assay (IRMA).

CONTACTS AND LOCATIONS:
Locations (1):
- Marwa Shafiek Saleh, Giza, Egypt